CLINICAL TRIAL: NCT01020123
Title: A 4-month, Randomized, Double-blind, Placebo- and Active-Controlled, Multi-centre, Parallel-Group Study, With an Optional 2-month Extension, to Evaluate Efficacy, Safety and Tolerability of AZD1656 as Add-on Treatment to Metformin in Type 2 Diabetes Mellitus Patients
Brief Title: Evaluate Efficacy, Safety and Tolerability of AZD1656 as Add-on Treatment to Metformin in Type 2 Diabetes Mellitus (TD2M) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1020C00009
Record Dates: First submitted 2009-11-11; First posted 2009-11-25 (Estimated); Results first posted 2012-11-26 (Estimated); Last update posted 2012-11-26 (Estimated); Status verified 2012-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II Diabetes Mellitus; metformin; glipizide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656; Glipizide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 2 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 3 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 4 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 5 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo
- 7 (Active Comparator): Glipizide administered to 1 group of patients
  Interventions: Drug: Glipizide

INTERVENTIONS:
Drug: AZD1656 — Different doses of AZD1656 administered to 5 groups of patients
  Arms: 1; 2; 3; 4; 5
Drug: Placebo — AZD1656 placebo and glipizide placebo administered to 1 group of patients
  Arms: 6
Drug: Glipizide — Glipizide administered to 1 group of patients
  Arms: 7

SUMMARY:
The primary aim is to evaluate Efficacy, Safety and Tolerability of AZD1656 as Add-on Treatment to Metformin in TD2M Patients

ELIGIBILITY:
Inclusion Criteria:

* female of non-childbearing potential
* Treated with maximally tolerated dose of metformin (≥ 1500mg/day) for at least 10 weeks prior to enrolment.
* Patients with HbA1c ≥ 7.5 but ≤ 10% at enrolment visit (Visit 1) can enter cohort 1.Patients with HbA1c between >10 % and <12 % can enter the open-label arm with AZD1656 (cohort 2)

Exclusion Criteria:

* Significant cardiovascular event within the last 6 months prior to enrolment or heart failure New York Heart Association (NYHA) class III-IV.
* Impaired renal function in terms of GFR<60 ml/min, based on Modification of Diet in Renal Disease Study Group (MDRD) calculation.
* Use of warfarin or amiodarone within 3 months prior to enrolment (screening) and use of potent CYP450 inhibitors, eg, ketoconazole and/or macrolide antibiotics within 14 days before randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Johnsson, Study Director — AstraZeneca R&D Mölndal; John Wilding, DM FRCP, Principal Investigator — University Hospital Aintree
Locations (77):
- Chile (4):
  - Research Site, Temuco, Región de la Araucanía
  - Research Site, Brentwood, TN
  - Research Site, Santiago
  - Research Site, Temuco
- Germany (11):
  - Research Site, Dresden, Saxony
  - Research Site, Brentwood, TN
  - Research Site, Aschaffenburg
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, Görlitz
  - Research Site, Hamburg
  - Research Site, Lübeck
  - Research Site, Magdeburg
- Hungary (11):
  - Research Site, Saint Laurent, QC
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Szekszárd
  - Research Site, Szigetvár
  - Research Site, Zalaegerszeg
- Latvia (8):
  - Research Site, Brentwood, TN
  - Research Site, Daugavpils
  - Research Site, Jelgava
  - Research Site, Jēkabpils
  - Research Site, Limbaži
  - Research Site, Riga
  - Research Site, Talsi
  - Research Site, Valmiera
- Lithuania (2):
  - Research Site, Brentwood, TN
  - Research Site, Kaunas
- Mexico (10):
  - Research Site, Aguascalientes, Aguascalientes
  - Research Site, Zapopan, Jalisco
  - Research Site, Monterrey, Mexico
  - Research Site, Cuernavaca, Morelos
  - Research Site, Monterrey, Nuevo León
  - Research Site, Brentwood, TN
  - Research Site, Meridas, Yucatán
  - Research Site, Mérida, Yucatán
  - Research Site, Chiuahua
  - Research Site, San Luis Potosí City
- Peru (7):
  - Research Site, Lima, Lima Province
  - Research Site, Brentwood, TN
  - Research Site, Callao
  - Research Site, Lambayeque
  - Research Site, Lima
  - Research Site, Piura
  - Research Site, Trujillo
- Poland (5):
  - Research Site, Brentwood, TN
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Kutno
  - Research Site, Wroclaw
- Romania (7):
  - Research Site, Alba Iulia, Alba
  - Research Site, Tg Mures, Mureș County
  - Research Site, Brentwood, TN
  - Research Site, Galati
  - Research Site, Ploieşti
  - Research Site, Sibiu
  - Research Site, Timișoara
- Sweden (3):
  - Research Site, Brentwood, TN
  - Research Site, Huddinge
  - Research Site, Lund
- United Kingdom (9):
  - Research Site, Paignton, Devon
  - Research Site, Liverpool, Merseyside
  - Research Site, Saint Laurent, QC
  - Research Site, Cardiff
  - Research Site, Chorley
  - Research Site, Glasgow
  - Research Site, Stevenage
  - Research Site, West Bromwich
  - Research Site, West Lothian

RESULTS

PARTICIPANT FLOW:
Groups:
- Higher Dose: 20-200 mg AZD1656 add on to metformin, titrated dose
- Lower Dose: 10-140 mg AZD1656 add on to metformin, titrated dose
- 40 mg Fixed Dose: 40 mg AZD1656 add on to metformin, fixed dose
- 20 mg Fixed Dose: 20 mg AZD1656 add on to metformin, fixed dose
- Placebo: Placebo add on to metformin
- Glipizide: 5-20 mg Glipizide add on to metformin, titrated dose
- Open Label: Open label, 20-200 mg AZD1656 add on to metformin, titrated dose
Period: Main Period
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Started | 93 | 91 | 52 | 40 | 88 | 94 | 72
Completed | 76 | 77 | 44 | 33 | 77 | 83 | 61
Not Completed | 17 | 14 | 8 | 7 | 11 | 11 | 11
Not completed — Withdrawal by Subject | 6 | 5 | 3 | 1 | 6 | 3 | 2
Not completed — Eligibility Criteria not fullfilled | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 5 | 2 | 2 | 1 | 1 | 2 | 1
Not completed — Protocol Violation | 4 | 4 | 2 | 5 | 2 | 3 | 2
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Unclasified | 2 | 0 | 1 | 0 | 1 | 3 | 6
Period: Extention Period
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Started | 40 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 35 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 19 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 13 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 31 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 38 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.) | 19 (Not everyone accepted protocol amendment allowing to enter extension period or was asked to enter.)
Completed | 37 | 33 | 17 | 12 | 31 | 36 | 18
Not Completed | 3 | 2 | 2 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label | Total
Number analyzed (Participants) | 93 | 91 | 52 | 40 | 88 | 94 | 72 | 530
Age Continuous [Mean (Full Range); unit: Year] | 57.1 [34 to 81] | 57.1 [32 to 80] | 54.4 [23 to 77] | 57.4 [35 to 80] | 56.9 [30 to 75] | 57.1 [36 to 78] | 53.1 [20 to 69] | 56 [20 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 46 | 22 | 19 | 45 | 46 | 37 | 262
  Male | 46 | 45 | 30 | 21 | 43 | 48 | 35 | 268

OUTCOME MEASURES:

1. Primary Outcome: HbA1c: Change From Baseline to 4 Month
Description: AZD1656 is analyzed in a ANCOVA model (Glipized and Open Label is Not Included in the model), FAS Prior to Rescue
Time Frame: Baseline to 4th Month
Population: The population is FAS prior to rescue, using the LOCF values (see table 27 in CSR)
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 80 | 82 | 47 | 34 | 82
Percentage | -1.25 (-1.14) [-1.49 to -1.01] | -1.26 (-1.14) [-1.49 to -1.02] | -0.67 (-0.62) [-0.99 to -0.36] | -0.61 (-0.60) [-0.98 to -0.24] | -0.45 (NA) [-0.69 to -0.21]

2. Secondary Outcome: FPG: to Evaluate Change From Baseline to 4 Month, Compared With Placebo, FAS Prior to Rescue.
Description: AZD1656 is analyzed in a ANCOVA model (Glipized and Open Label is Not Included in the model), FAS Prior to Rescue.
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 29 in CSR)
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 90 | 87 | 49 | 39 | 85
mmol/L | -0.818 (-1.373) [-1.331 to -0.304] | -1.08 (-1.642) [-1.603 to -0.558] | 0.041 (-0.652) [-0.656 to 0.738] | 0.024 (-0.737) [-0.757 to 0.804] | -0.182 (NA) [-0.71 to 0.347]

3. Secondary Outcome: SMPG: Change From Baseline to 4 Month, Compared With Placebo, FAS Prior to Rescue.
Description: AZD1656 is analyzed in a ANCOVA model (Glipized and Open Label is Not Included in the model), FAS Prior to Rescue.
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 31 in CSR)
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 58 | 63 | 38 | 26 | 57
mmol/L | -1.596 (-2.206) [-2.176 to -1.016] | -1.557 (-2.155) [-2.117 to -0.997] | -0.874 (-1.586) [-1.591 to -0.157] | -0.604 (-1.437) [-1.472 to 0.265] | -0.213 (NA) [-0.799 to 0.372]

4. Secondary Outcome: OGTT/Plasma Glucose
Description: The relative change in AUC
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 142 in CSR)The first 50% of patients enrolled in the study were supposed to undertake OGTT, actual number participating was 52%. However, more than 60% of the OGTT patients were excluded from the analyses, as their measurements did not comply with the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 17 | 13 | 7 | 8 | 17
ratio | 0.92 [0.82 to 1.02] | 0.84 [0.75 to 0.96] | 1.02 [0.86 to 1.22] | 0.99 [0.84 to 1.16] | 0.99 [0.88 to 1.10]

5. Secondary Outcome: OGTT/Insulin
Description: The Relative Change in AUC FAS Prior to Rescue
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 146 in CSR)The first 50% of patients enrolled in the study were supposed to undertake OGTT, actual number participating was 52%. However, more than 60% of the OGTT patients were excluded from the analyses, as their measurements did not comply with the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 16 | 12 | 6 | 10 | 16
ratio | 0.81 [0.66 to 0.99] | 1.08 [0.85 to 1.36] | 0.97 [0.69 to 1.35] | 0.90 [0.69 to 1.16] | 0.91 [0.74 to 1.12]

6. Secondary Outcome: OGTT/C-peptide
Description: The relative change, FAS prior to rescue
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 150 in CSR)The first 50% of patients enrolled in the study were supposed to undertake OGTT, actual number participating was 52%. However, more than 60% of the OGTT patients were excluded from the analyses, as their measurements did not comply with the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 17 | 13 | 7 | 10 | 16
ratio | 0.97 [0.85 to 1.10] | 1.11 [0.96 to 1.29] | 0.90 [0.74 to 1.10] | 0.95 [0.81 to 1.13] | 1.00 [0.87 to 1.14]

7. Secondary Outcome: OGTT/Pro-insulin/Insulin
Description: The relative change, FAS prior to rescue
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the LOCF values (see table 154 in CSR)The first 50% of patients enrolled in the study were supposed to undertake OGTT, actual number participating was 52%. However, more than 60% of the OGTT patients were excluded from the analyses, as their measurements did not comply with the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 16 | 12 | 6 | 10 | 14
Ratio | 1.496 [1.250 to 1.791] | 1.199 [0.973 to 1.476] | 1.248 [0.932 to 1.672] | 1.431 [1.135 to 1.805] | 1.185 [0.979 to 1.436]

8. Secondary Outcome: HbA1c ≤ 7
Description: Number of responders ≤ 7, FAS prior to rescue.
Time Frame: baseline to 4 month
Population: The population is FAS prior to rescue, using the observed cases (see table 35 in CSR).
Measure: Number; unit: Participants
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 74 | 73 | 38 | 32 | 69 | 78 | 48
Participants | 43 | 43 | 14 | 11 | 16 | 50 | 24

9. Secondary Outcome: HbA1c ≤ 6.5
Description: Number of Responders ≤ 6.5, FAS Prior to Rescue
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 228 in CSR).
Measure: Number; unit: Participants
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 74 | 73 | 38 | 32 | 69 | 78 | 48
Participants | 35 | 27 | 9 | 4 | 9 | 30 | 16

10. Secondary Outcome: LDL-C: Mean Ratio
Description: Geometric mean ratio (safety analysis set, regardless of rescue) and a 95 % CI.
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 228 in CSR)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 74 | 75 | 43 | 33 | 73
ratio | 1.07 (29.5) [1.01 to 1.13] | 1.02 (20.6) [0.97 to 1.08] | 1.07 (38.5) [0.99 to 1.15] | 1.04 (23.1) [0.96 to 1.13] | 1.02 (19.3) [0.97 to 1.08]

11. Secondary Outcome: HDL-C: Change From Baseline
Description: Geometric mean ratio (safety analysis set, regardless of rescue) and a 95 % CI.
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 230 in CSR)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 75 | 76 | 43 | 33 | 74
ratio | 1.06 (6.2) [1.02 to 1.09] | 1.06 (5.1) [1.03 to 1.10] | 1.05 (7.8) [1.01 to 1.09] | 1.03 (4.1) [0.99 to 1.08] | 1.03 (5.3) [1.00 to 1.06]

12. Secondary Outcome: Total Cholesterol: Change From Baseline
Description: Geometric mean ratio (safety analysis set, regardless of rescue) and a 95 % CI.
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 232 in CSR)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 75 | 76 | 43 | 33 | 74
ratio | 1.09 (36.9) [1.04 to 1.13] | 1.08 (60.2) [1.04 to 1.12] | 1.07 (41.6) [1.02 to 1.13] | 1.04 (25.3) [0.98 to 1.10] | 1.03 (26.0) [0.99 to 1.07]

13. Secondary Outcome: Triglycerides: Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 226 in CSR)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 75 | 43 | 33 | 74 | 82 | 58
mg/dL | 40.9 (115.3) [39.2 to 114.4] | 38.7 (99.3) [38.7 to 99.3] | 19.8 (185.3) [19.8 to 185.3] | 4.4 (49.3) [4.4 to 49.3] | 13.7 (139.4) [13.4 to 139.4] | 18.7 (152.8) [13.7 to 139.4] | 29.8 (174.3) [18.7 to 152.8]

14. Secondary Outcome: C-reactive Protein: Change From Baseline
Description: Geometric mean ratio (safety analysis set, regardless of rescue) and a 95 % CI
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 234 in CSR)
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo
Number analyzed (Participants) | 75 | 76 | 43 | 33 | 75
ratio | 0.30 (0.88) [0.08 to 0.52] | 0.08 (0.86) [-0.14 to 0.30] | 0.09 (0.99) [-0.20 to 0.30] | 0.06 (0.74) [-0.40 to 0.27] | -0.02 (0.75) [-0.24 to 0.20]

15. Secondary Outcome: Systolic Blood Pressure, Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 237 in CSR)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 73 | 38 | 32 | 69 | 79 | 58
mmHg | -0.4 (12.6) | 0.4 (9.9) | 5.7 (11.3) | 0.1 (12.6) | -0.2 (13.7) | -1.1 (13.5) | -0.3 (11.7)

16. Secondary Outcome: Diastolic Blood Pressure, Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 240 in CSR)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 73 | 38 | 32 | 69 | 79 | 58
mmHg | 1.1 (8.6) | 1.4 (8.5) | 1.3 (9.1) | -0.9 (10.8) | -0.3 (8.5) | -0.1 (7.2) | 0.5 (7.7)

17. Secondary Outcome: Pulse, Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 236 in CSR)
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 73 | 38 | 32 | 69 | 79 | 58
Beats/min | 0.4 (8.8) | 1.6 (7.9) | 1.3 (7.9) | 0.3 (9.1) | -1.1 (9.4) | -0.4 (11.6) | 1.3 (8.5)

18. Secondary Outcome: Weight, Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 244 in CSR)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 73 | 38 | 32 | 69 | 79 | 48
kg | -0.3 (2.5) | -0.6 (2.9) | -1.2 (2.7) | -1.4 (2.3) | -1.0 (2.5) | 1.0 (3.4) | -0.4 (4.4)

19. Secondary Outcome: QTcF; Electorcardiagram Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 258 in CSR)
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 74 | 76 | 43 | 34 | 77 | 83 | 63
msec | 4.4 (15.6) | 4.0 (14.5) | -2.6 (12.6) | 3.8 (17.9) | 2.2 (13.8) | 2.7 (21.5) | 1.6 (16.4)

20. Secondary Outcome: Haemoglobin; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: population is safety analysis set regardless of rescue, using the observed cases (see table 197 in CSR)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 76 | 77 | 44 | 32 | 76 | 83 | 61
g/dL | -0.20 (0.68) | -0.18 (0.62) | 0.00 (0.63) | -0.11 (0.69) | -0.20 (0.71) | 0.02 (0.69) | -0.25 (0.76)

21. Secondary Outcome: Leukocytes; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 198 in CSR)
Measure: Mean (Standard Deviation); unit: *10^3 cells/µL
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 76 | 77 | 44 | 32 | 76 | 83 | 61
*10^3 cells/µL | 0.39 (1.29) | 0.34 (1.59) | 0.35 (1.41) | -0.15 (1.09) | -0.8 (1.09) | 0.27 (1.43) | -40 (1.31)

22. Secondary Outcome: Sodium; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 215 in CSR)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 77 | 44 | 33 | 76 | 83 | 60
mEq/L | -0.6 (2.4) | -0.7 (2.4) | -0.4 (3.0) | -0.1 (2.6) | 0.0 (2.6) | -0.6 (3.3) | 0.5 (2.6)

23. Secondary Outcome: Potassium; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 214 in CSR)
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 77 | 43 | 32 | 75 | 82 | 58
mEq/L | 0.02 (0.45) | -0.02 (0.26) | 0.00 (0.35) | -0.01 (0.29) | -0.02 (0.34) | 0.07 (0.39) | 0.05 (0.38)

24. Secondary Outcome: Creatinine; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 211 in CSR)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 77 | 43 | 32 | 75 | 82 | 59
IU/L | 0.4 (70.5) | -9.9 (87.8) | 8.5 (88.7) | -8.3 (39.1) | -0.1 (32.2) | 15.9 (67.1) | -7.3 (47)

25. Secondary Outcome: ALT; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 206 in CSR)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 76 | 43 | 32 | 75 | 82 | 59
IU/L | 2.0 (12.0) | 1.7 (14.8) | 3.2 (17.7) | -1.8 (-1.8) | -0.4 (11.3) | 2.0 (15.3) | -0.4 (15.5)

26. Secondary Outcome: AST; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 207 in CSR)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 76 | 43 | 32 | 75 | 82 | 59
IU/L | 2.4 (9.8) | 2.0 (11.0) | 2.8 (13.1) | -0.6 (8.9) | -0.1 (7.9) | 2.1 (13.3) | 2.7 (9.6)

27. Secondary Outcome: Alkaline Phosphatase; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 208 in CSR)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 77 | 44 | 33 | 76 | 83 | 59
IU/L | 3.8 (17.5) | -1.3 (13.3) | 0.0 (13.6) | -1.8 (11.9) | -3.4 (11.5) | -4.2 (16.7) | -11.7 (24.7)

28. Secondary Outcome: Bilirubin; Change From Baseline
Description: Summary statistic of change from baseline
Time Frame: baseline to 4 month
Population: The population is safety analysis set regardless of rescue, using the observed cases (see table 209 in CSR)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Number analyzed (Participants) | 75 | 77 | 44 | 33 | 76 | 83 | 59
mg/dL | -0.02 (0.17) | -0.06 (0.21) | 0.02 (0.13) | -0.05 (0.20) | -0.01 (0.20) | -0.07 (0.20) | -11.7 (24.7)

29. Secondary Outcome: CL/F to Characterise the PK Properties of AZD1656.
Description: The value is calculated using an allometric model (of a patient weighting 75 kg). The value is independent treatment given.
Time Frame: at 4 month
Measure: Mean (Standard Error); unit: L/h
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Open Label
Number analyzed (Participants) | 86 | 87 | 49 | 39 | 70
L/h | 9.29 (3.7) | 9.29 (3.7) | 9.29 (3.7) | 9.29 (3.7) | 9.29 (3.7)

30. Secondary Outcome: EC50 to Characterise the PD Properties of AZD1656.
Description: The value is model based. The value is independent treatment given.
Time Frame: at 4 month
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Open Label
Number analyzed (Participants) | 86 | 87 | 49 | 39 | 70
nmol/L | 60.2 (14) | 60.2 (14) | 60.1 (14) | 60.2 (14) | 60.2 (14)

ADVERSE EVENTS:
Time Frame: Baseline - 6 month
Description: Safety was collected in 6 month
Arm/Group | Higher Dose | Lower Dose | 40 mg Fixed Dose | 20 mg Fixed Dose | Placebo | Glipizide | Open Label
Serious Adverse Events (participants affected / at risk) | 2/92 | 1/90 | 1/50 | 1/40 | 2/87 | 3/93 | 1/71
Other Adverse Events (participants affected / at risk) | 22/92 | 36/90 | 20/50 | 10/40 | 14/87 | 35/93 | 9/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Higher Dose (N=92) | Lower Dose (N=90) | 40 mg Fixed Dose (N=50) | 20 mg Fixed Dose (N=40) | Placebo (N=87) | Glipizide (N=93) | Open Label (N=71)
Angina Unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failur acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose (N=92) | Lower Dose (N=90) | 40 mg Fixed Dose (N=50) | 20 mg Fixed Dose (N=40) | Placebo (N=87) | Glipizide (N=93) | Open Label (N=71)
Nasopharyngitis (Infections and infestations) | 4 | 9 | 2 | 1 | 6 | 3 | 3 — This iformation is based on tables 182 and 183 in the CSR
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 2 | 2 | 0 | 0 — This iformation is based on tables 182 and 183 in the CSR
Diarrhoea (Gastrointestinal disorders) | 4 | 7 | 3 | 3 | 3 | 3 | 0 — This iformation is based on tables 182 and 183 in the CSR
Nausea (Gastrointestinal disorders) | 2 | 2 | 4 | 0 | 1 | 1 | 1 — This iformation is based on tables 182 and 183 in the CSR
Vomiting (Gastrointestinal disorders) | 0 | 2 | 5 | 0 | 0 | 1 | 0 — This iformation is based on tables 182 and 183 in the CSR
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 0 | 2 | 0 — This iformation is based on tables 182 and 183 in the CSR
Asthenia (General disorders) | 2 | 4 | 1 | 0 | 0 | 7 | 0 — This iformation is based on tables 182 and 183 in the CSR
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 4 | 1 | 1 | 0 | 10 | 2 — This iformation is based on tables 182 and 183 in the CSR
Tremor (Nervous system disorders) | 4 | 4 | 1 | 1 | 0 | 10 | 1 — This iformation is based on tables 182 and 183 in the CSR
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 0 | 2 | 6 | 2 — This iformation is based on tables 182 and 183 in the CSR

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less